CLINICAL TRIAL: NCT05665764
Title: Enhancing Precision Sleep Medicine in Traumatic Brain Injury: Examining the Feasibility of Home-Based Measurement of Circadian Timing
Brief Title: The Feasibility of Home-Based Measurement of Circadian Timing for Veterans With TBI and Insomnia
Acronym: Home DLMO
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: D4414-P
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Brain Injuries, Traumatic; Sleep Initiation and Maintenance Disorders
Keywords: Circadian phase; Veteran; Traumatic Brain Injury; Insomnia
MeSH Terms: conditions — Brain Injuries, Traumatic; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens will be retained. Saliva samples will be collected and tested for dim light melatonin onset as part of the study, after which they will be destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Veterans: Veterans will be the primary cohort for this study. Veterans who will be enrolled with have current insomnia and a history of traumatic brain injury.
- Caregivers: Caregivers of enrolled veterans will be an optional cohort for this study. If applicable and willing to participate, caregivers of enrolled Veterans will be asked to provide collateral information regarding the Veteran's experience with the study.

SUMMARY:
Veterans with traumatic brain injury (TBI) frequently experience insomnia, which is linked with delayed TBI recovery, more severe functional impairment, and exacerbation of disabling TBI after-effects such as depression, chronic pain, and fatigue. Current research suggests that TBI can impact numerous systems involved in sleep, suggesting that insomnia can have various causes and that a "one-size-fits-all" approach to treatment is likely inadequate. As such, it is necessary to determine which Veterans may benefit from standard evidence-based treatments, such as Cognitive Behavior Therapy for Insomnia, and which may require enhanced treatments targeting specific underlying mechanisms.

An emerging body of evidence has established a link between circadian rhythm disruption and post-TBI insomnia. A mismatch between circadian and desired sleep timing (i.e., "circadian misalignment") is common following TBI, as evidenced by disruptions of key circadian rhythms involved in sleep regulation (e.g., melatonin production), as well as the onset of circadian rhythm sleep-wake disorders. Importantly, circadian-driven sleep disturbances require specialized treatments that target circadian rhythms (i.e., "chronotherapies"), such as timed sleep windows or enhanced light exposure, as standard treatment approaches can fail to address or even exacerbate the underlying circadian misalignment. Thus, circadian misalignment represents a novel and modifiable treatment target and has the potential to improve functional outcomes in Veterans with TBI and insomnia.

Detection of circadian misalignment and optimal use of chronotherapies require the ability to measure circadian phase (i.e., timing of the central circadian clock). However, current sleep medicine in TBI is hampered by a lack of pragmatic options for measuring circadian phase. This is because laboratory dim light melatonin onset (DLMO), the gold standard measure of circadian phase, is time and cost prohibitive, requiring specialized sample (e.g., saliva) collection facilities and placing substantial burden on the patient. Recently, novel methods of DLMO measurement have been developed that may enhance the accessibility and practicality of circadian phase assessment, although, as of yet, they have not been used in Veterans with TBI. The proposed single-arm, longitudinal study seeks to evaluate the feasibility of two methods of measuring DLMO in the home environment of Veterans with TBI and insomnia: 1) direct measurement of self-collected salivary melatonin; and 2) indirect estimation of DLMO using activity and light-exposure data collected through actigraphy. Additionally, this study seeks to explore the relationships between circadian misalignment, sleep disturbance, and functional impairment in Veterans with TBI.

The specific aims of this study are to: Aim 1) evaluate the feasibility of two methods of home DLMO measurement (i.e., self-collected salivary melatonin and actigraphy data) in Veterans with TBI and insomnia; and Aim 2) examine associations between circadian misalignment (i.e., the difference in timing between DLMO and attempted sleep onset), sleep disturbance, and functional impairment. Veterans with TBI and insomnia will be asked to wear a wrist-based actigraphy device for one week, which will collect data on light exposure and sleep-wake states. They will then be asked to self-collect seven hourly saliva samples under dim light conditions in their own home and mail them to a testing facility using a provided pre-paid shipping label. Saliva samples will be used to directly measure DLMO and actigraphy data will be used to indirectly estimate DLMO using established mathematical models of the human circadian pacemaker. Evaluating the feasibility of home DLMO measurement is a crucial first step for enhancing precision sleep medicine for Veterans with TBI and insomnia. Findings will inform the development and testing of tailored sleep interventions for use with this patient population.

DETAILED DESCRIPTION:
Background and Significance:

Insomnia is a pervasive problem among Veterans with traumatic brain injury (TBI). Veterans with TBI frequently experience sleep disturbances following their injury. Insomnia, an impairing disorder characterized by difficulty initiating or maintaining sleep, is the most common sleep disturbance reported following TBI. Indeed, Veterans with TBI are 50% more likely to develop future insomnia compared to their non-injured peers.

The development of insomnia following TBI can delay recovery and contribute to functional impairments. Compared to TBI patients with normal sleep, those with insomnia have up to eightfold greater odds of functional impairment in the six months after injury. Post-TBI, United States (U.S.) Veterans who had poor sleep were more likely to report pain was interfering with their lives, have diminished health-related quality of life, and perform worse on neurobehavioral measures. A large-sample study found that insomnia was associated with decreased life satisfaction both immediately following TBI and one-year post-injury. Furthermore, insomnia is strongly associated with, and can exacerbate, other TBI sequelae such as depression, chronic pain, and fatigue, which can further delay rehabilitation and recovery from TBI.

Mechanisms underlying insomnia in TBI are heterogeneous, indicating that a "one-size-fits-all" approach to treatment is likely inadequate. While the precise mechanisms that underlie insomnia after TBI remain unknown, the extant research suggests that TBI can impact numerous systems that regulate sleep and wake states. Insomnia can result from damage to specific brain regions involved in sleep initiation (e.g., basal forebrain). Widespread brain damage, such as diffuse axonal injury, can disturb sleep through disruption of neuronal signaling, buildup of cellular waste byproducts, and toxic metabolic cascades. Perturbation of hormonal systems are also associated with insomnia following brain injury. Moreover, physical and psychological sequelae of TBI, such as pain, depression, or posttraumatic stress disorder (PTSD), can contribute to insomnia. Therefore, it is necessary to differentiate Veterans who may benefit from standard evidence-based treatments, such as Cognitive Behavioral Therapy for Insomnia (CBTI), and those who may require enhanced treatments targeting specific underlying mechanisms.

One distinct, but understudied, causal mechanism implicated in post-TBI insomnia is disruption to the circadian system. Circadian rhythms are changes in biochemical, physiological, or behavioral processes that repeat over the course of approximately 24 hours and are responsive to external cues such as light exposure. A mismatch between circadian and desired sleep timing (i.e., "circadian misalignment") can disturb sleep, manifesting as insomnia or circadian rhythm sleep-wake disorders (CRSDs) like delayed or advanced sleep phase disorders. Following TBI, circadian misalignment is common, as seen in perturbations of key circadian rhythms involved in sleep regulation (e.g., melatonin production), as well as the manifestation of CSRDs. This may be because TBI dysregulates the expression of circadian clock genes, which in turn is correlated with disruption of day/night activity rhythms. Another potential pathway linking TBI to circadian misalignment is the immune system, which communicates bidirectionally with the circadian system and is activated following TBI. Post-TBI inflammation may induce circadian desynchrony-a lack of temporal coordination across tissues, organs, and molecular processes-thus impairing homeostatic control and driving a pathological feedback loop of further inflammation, circadian misalignment, and resulting sequelae. Indeed, many impairments that arise from TBI, including sleep-wake disturbances, are also observed in cases of circadian desynchronization, further implicating circadian misalignment in TBI symptomatology.

Accurate detection, and subsequent correction, of circadian misalignment represents a unique, novel, and modifiable treatment target that has the potential to improve the efficacy of circadian-targeted treatments ("chronotherapies") and functional outcomes for Veterans with TBI and insomnia. Failure to detect circadian misalignment underlying insomnia can lead to a choice of an ineffective intervention. Treating circadian-driven sleep disturbances requires specialized treatment approaches, such as timed exposure to light and darkness or melatonin supplementation, that aim to modify the timing or signaling strength of the individual's internal biological clock. By acting upon this clock, chronotherapies can adjust the timing of sleep-wake cycles and consolidate irregular or fragmented sleep. However, appropriate and efficacious administration of chronotherapies requires an understanding of the precise timing of the individual's biological clock (i.e., circadian phase), as the potency of these interventions vary across the internal day and night and can range from salubrious to ineffective or even harmful. For example, when unguided by circadian phase, standard sleep interventions, like sleep restriction therapy (the main component of CBTI), may fail to address underlying circadian misalignment or may even exacerbate it. Additionally, the degree of side effects associated with acute sleep restriction, such as impaired attention, daytime sleepiness, disrupted mood, and dysregulated autonomic function, depend upon the individual's circadian phase prior to the start of the intervention. Thus, accurate measurement of circadian misalignment would not only allow providers to identify when an empirically supported chronotherapy (alone or in combination with other sleep interventions) may be indicated, but it could also help providers optimize the delivery of chronotherapies for insomnia and monitor changes to circadian phase, thereby improving treatment response.

Sleep medicine for TBI is hampered by a lack of pragmatic options for measuring circadian phase. Time of dim light melatonin onset (DLMO) is currently considered the "gold standard" for measuring circadian phase and is an important tool for identifying circadian misalignment in insomnia. However, laboratory measurement of DLMO is time and cost prohibitive, as patients must report to the collection facility 6-8 hours before their typical bedtime, remain in supervised dim-light conditions, and give frequent samples (e.g., saliva) until their bedtime or later. Such requirements make the routine measurement of DLMO in clinical settings impractical. Indeed, lack of testing for objective markers of circadian phase like DLMO has been recently highlighted as a significant gap in the identification of circadian misalignment when diagnosing and treating sleep disorders. Alternatives to laboratory DLMO that allow healthcare providers to pragmatically and accurately measure circadian phase are needed to advance precision sleep medicine in TBI.

Novel methods of DLMO measurement have been developed that may enhance the accessibility and practicality of circadian phase assessment; however, their feasibility for Veterans with TBI and insomnia remains unknown. In the past decade, two new approaches for measuring DLMO at home have emerged. The first involves directly testing for DLMO in self-collected saliva samples. Although similar to laboratory DLMO measurement, in that Veterans are still required to collect frequent saliva samples under dim light conditions, self-collected saliva allows Veterans to remain in the comfort of their own homes during the collection procedures. This approach could increase uptake of DLMO measurement by clinicians, as it would circumvent the need for a referral to another facility or service. Initial research has shown that obtaining DLMO from self-collected saliva is viable for over 85% of participants, suggesting that patients are able to adhere to collection procedures. The second novel approach involves indirectly measuring DLMO from the patient's daily activity levels and light exposure. By employing established mathematical models of the human circadian pacemaker, DLMO can be estimated based on the amount and timing of light exposure throughout the day, as well as the timing of sleep. Excitingly, the data needed for indirect DLMO measurement can be acquired passively via wearable sensor technology, such as a wrist-worn actigraphy device, meaning that circadian phase can be assessed with minimal patient burden. Previous research has achieved high rates of data acquisition using this approach and successfully estimated DLMO with as little as a few days of actigraphy data. More important, both home DLMO approaches have been validated against laboratory DLMO in healthy participants and participants with disordered sleep, suggesting that they can measure circadian phase with enough accuracy to be used in clinical practice.

While these initial findings are promising, additional work is needed before they can be applied to the care of insomnia in Veterans with TBI. Potential barriers inherent to each home DLMO method may limit successful measurement of circadian phase. For example, the requirements of home saliva collection, such as avoiding light exposure and providing samples at prespecified times, may be difficult for Veterans experiencing TBI symptoms like cognitive impairment. Similar difficulties may be encountered when using actigraphy, as Veterans may inadvertently cover the light sensor with clothing or forget to wear the device continuously over the assessment period. Establishing the feasibility of home DLMO methods in Veterans with TBI and insomnia is a vital first step for their implementation in clinical care.

Significance. In summary, there is a crucial need for circadian phase assessment to be made a routine part of insomnia care for Veterans with TBI, yet the primary way of doing so, laboratory DLMO, is rarely used due to its high level of burden. This project will address the above gap by evaluating the feasibility of two pragmatic methods for measuring circadian phase via DLMO in the home environment: direct measurement of DLMO through self-collected saliva and indirect measurement of DLMO via activity and light exposure data. Additionally, this study will be the first direct exploration of the hypothesized relationships between circadian misalignment, functional impairment, and sleep disturbance in Veterans with TBI. Thus, findings from this study may inform the development and testing of tailored sleep interventions for Veterans with TBI, with the goal of enhancing functional outcomes by restoring synchrony between biological timing and psychosocial demands. For example, accurate and accessible measurement of circadian phase will allow providers to: 1) detect underlying circadian misalignment in insomnia that would otherwise go unnoticed; 2) provide Veterans with TBI with an appropriate evidence-based sleep intervention (i.e., chronotherapy or standard care); and 3) monitor treatment response and adjust accordingly. Finally, this research has broad implications for a range of populations seeking rehabilitative care, including those with a history of stroke, spinal cord injury, and serious mental illness.

Description of Population to be Enrolled:

Potential participants will be all willing and eligible U.S. military Veterans aged 18-64 from the following populations: 1) those seeking outpatient services at the Rocky Mountain Regional Veterans Affairs (VA) Medical Center; and 2) those in existing clinical and research databases (e.g., the Rocky Mountain Mental Illness Research, Education and Clinical Center [RM MIRECC] research database).

Study Design and Research Methods:

Recruitment. Multiple means will be used to inform potential participants (i.e., Veterans with TBI and insomnia receiving care in the Veterans Health Administration) about this research project. This includes letters, flyers, social media, advertisements, presentations, and/or involving professionals treating Veterans. The RM MIRECC recruitment team will assist.

Screening. A research team member will explain the procedures to interested participants (via phone or video conference) and complete the screening checklist. If applicable, primary caregivers will be invited to attend screening and subsequent sessions. Those who pass screening will be scheduled for in-person eligibility evaluation and Consent/Baseline.

Eligibility, Consent, and Baseline Assessment. Informed consent will be obtained from interested participants who pass the initial screening (and caregivers, if applicable, to obtain collateral data). Eligibility criteria will be established via administration of the OSU TBI-ID, SCISD-R, and SCID. Following confirmation of eligibility, a member of the research team will administer other measures via the Research Electronic Data Capture (REDCap) survey system. Actigraphy and home saliva collection dates will be scheduled. At this time, a Preparation call will also be scheduled to take place the day before saliva collection.

Practice Training Session. Following baseline assessment (during the same visit), a practice session will take place, so the participant can learn to use the actigraphy device and the home saliva collection kit (Salimetrics, CA, USA), both of which will be given to the participant at the end of the session along with instructional handouts. At the end of the practice session, a brief skills check (e.g., simulating saliva collection procedures) will be conducted to address any remaining difficulties in understanding the study tasks. Furthermore, the practice session will be piloted with the first four study participants and adjustments to the protocol will be made as needed. A step-by-step video on how to complete saliva collection will also be created for this study and hosted on a study website. Based on study findings, teaching resources will be made public for use by other clinicians and researchers. Participants will be provided with locations of return FedEx facilities (for returning saliva samples) closest to their home. Time to complete Baseline procedures and the practice session will be 2.5 hours.

Collection of Actigraphy and Sleep Diaries. For the week prior to their home salivary melatonin collection, participants will be asked to wear an actigraphy device continuously on their non-dominant wrist. They will be instructed to leave the device uncovered, such as by clothing, to allow the light sensor to function properly. Participants will also be asked to complete a daily sleep diary (5 minutes). They will receive a REDCap email link each morning for electronic data submission. A research team member will provide instructions on how to enter sleep diary data. During the week of sleep diary collection, participants will receive follow-up reminders (either by phone or email) if diary responses are not entered during the day. Participants will not be required to change their daily routines in any other way.

Home Saliva Collection. Pre-collection/Preparation Appointment. The day before saliva collection, participants will be called to remind them of the process. The research team member will go over each step, ensure participants have the correct collection times recorded, and answer any questions. The saliva kit contains all necessary materials for the storage and shipping of specimens (e.g., 7 pre-labeled cryovials). Along with the saliva kit, participants will be provided with a nightlight to facilitate collection, as well as a handout to guide them through the collection process based on the Salimetrics DLMO Profile Saliva Collection protocol. Participants will be asked to avoid alcohol and caffeine for 24 hours prior to saliva collection and to avoid pitted fruit and bananas during the day of collection. The provided handout will also include self-reported checks for methods adherence (e.g., avoiding food, caffeine), which will supplement the objective light adherence check (see next section).

Collection Day. At 5.5 hours prior to their typical self-reported bedtime, participants will be asked to reduce all sources of light as much as possible. Participants will be asked to remain in dim light (e.g., 40-watt lightbulb exposure or lower, closed blinds) and to reduce all electronic screen brightness as much as possible during the saliva collection process, as light exposure can inhibit melatonin production. The nightlight will be provided to assist in dimming the home. As an adherence check, light exposure during saliva collection will continue to be measured using the already provided actigraphy device. Participants will also be asked to refrain from napping, eating major meals, or brushing teeth during the collection period but will be allowed to consume light snacks. Saliva collection will then begin 5 hours prior to the participant's typical bedtime. Collection will take place each hour until 7 samples have been obtained (5 hours prior to bedtime until 1 hour after typical bedtime). For the 10 minutes prior to each collection, participants will be asked to refrain from eating any food or drinks other than water and to rinse their mouths with water. At the collection time, participants will be asked to provide passive drool using the labeled cryovial and record the collection time. They will be asked to store each saliva sample in the fridge or freezer when actively collecting saliva and then store all saliva samples in the freezer once collection is finished, until they are ready to drop the samples off at a FedEx shipping location for overnight shipping using the prepared shipping label. At this point, participants will also return the actigraphy device either in person or via a prepared shipping label. DLMO timing will be determined by Salimetrics laboratory services.

Qualitative Interview. A brief qualitative interview will be administered to participants (and caregivers, when applicable), including those who discontinue the study early (if possible). This will provide data regarding user experience with the DLMO methods, including potential facilitators and barriers.

Data Analysis Plan:

Aim 1. Each home DLMO measurement method will be evaluated separately and considered feasible if 70% participants provide adequate data for measurement of DLMO.

Aim 2. Linear regressions will be conducted to explore the association between circadian misalignment (independent variable) and either functional impairment or sleep disturbance (dependent variables). Functional impairment will be assessed using the WHODAS 2.0 summary score. Sleep disturbance will be assessed using the PROMIS sleep disturbance total score. Circadian misalignment will be defined as the difference in time between DLMO and the average sleep diary-based bedtime. Values for circadian misalignment will be calculated for each home DLMO method and evaluated in four separate statistical models. Covariates for all models will include age, gender, depressive symptom severity, and PTSD symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* History of traumatic brain injury
* Current insomnia

Exclusion Criteria:

* Alcohol or substance abuse in the past 12 months
* History of psychotic or bipolar disorders
* Currently using of beta-blockers or melatonin-related substances (including over-the-counter or herbal products)
* Currently participating in a sleep-targeted psychotherapy
* Transmeridian travel (i.e., change in at least 2 time zones) in the past month
* Shift work (i.e., at least 6 hours between 10 pm and 8 am) in the past 6 months
* Currently pregnant or lactating
* Current untreated sleep apnea
* Lack of access to a home freezer
* Blindness
* Inability to independently provide informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potential participants will be all willing and eligible U.S. military Veterans aged 18-64 from the following populations: 1) those seeking outpatient services at the Rocky Mountain Regional Veterans Affairs (VA) Medical Center; and 2) those in existing clinical and research databases (e.g., the Rocky Mountain Mental Illness Research, Education and Clinical Center [RM MIRECC] research database).
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of Home Dim Light Melatonin Onset (Self-Collected Saliva) | One week
  This outcome will be considered feasible if 70% participants provide adequate data for measurement of dim light melatonin onset (DLMO). For the self-collected salivary DLMO method, adequate data will entail: 1) collection and return of at least 5 saliva samples; 2) <5 minutes discrepancy between the reported and pre-specified collection times for the two saliva samples ultimately used to establish DLMO; and 3) 50 lux of light exposure within 30 minutes of the two saliva samples ultimately used to establish DLMO.
Feasibility of Home Dim Light Melatonin Onset (Actigraphy) | One week
  This outcome will be considered feasible if 70% participants provide adequate data for measurement of dim light melatonin onset (DLMO). For the actigraphy DLMO method, adequate data will entail wearing the actigraphy device for at least 2 continuous days, with no interval of missing data (e.g., from covering the light sensor) during that time greater than 2 consecutive hours.

SECONDARY OUTCOMES:
Functional Impairment (WHODAS 2.0 Summary Score) | Baseline
  WHO Disability Assessment Schedule 2.0 (WHODAS 2.0). The WHODAS 2.0 is a reliable and valid assessment for health and disability that spans six domains of functioning, including cognition, mobility, self-care, interactions with others, life activities, and participation in community activities.
Sleep Disturbance (PROMIS Sleep Disturbance Total Score) | Baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance. The PROMIS sleep disturbance is a 27-item self-report measure with excellent psychometric properties that assesses perceptions of sleep quality and sleep disturbance.

OTHER OUTCOMES:
Circadian Misalignment (Salivary Dim Light Melatonin Onset) | One week
  The difference in timing between dim light melatonin onset measured by self-collected saliva and the average sleep diary-based bedtime.
Circadian Misalignment (Actigraphy Dim Light Melatonin Onset) | One week
  The difference in timing between dim light melatonin onset measured by actigraphy and the average sleep diary-based bedtime.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Reis, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Final, deidentified, and anonymous data used in publications following this study will be made available upon request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data used for publications may be made available until data are destroyed per institutional requirements.
Access Criteria: Data will be made available for the validation of published findings or to support exploration of novel hypotheses. Requests to use data will be subject to a formal approval process. If approved, the requestor will be required to complete a data use agreement.

DOCUMENTS (1):
  • Informed Consent Form (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT05665764/ICF_000.pdf